| Official Title: | PROMOTE Pilot Study: Pharmacy Multimodal |
|-----------------|---------------------------------------------------|
| | Communication Strategy to Promote HPV Vaccination |
| NCT Number: | NCT04660331 |
| Document Type: | Informed Consent Form |
| Date of the | December 05, 2022 |
| Document: | |

#### V. 11/10/2022 CTMS# RG1007825, IR# 10600

## PROMOTE Pilot Study Pharmacy Staff Aim 2 Online Consent Form

Email subject line: Invitation to join the PROMOTE Pilot Study

Re: Promote Pilot Study Pharmacy Staff Online Consent Form

Hello,

We are writing to invite you to participate in a research study that seeks to understand the perspectives of pharmacy staff on delivering HPV vaccinations for children 9-17 years old in pharmacies.

The study is called "PROMOTE Pilot Study: Pharmacy multimodal communication strategy to promote HPV vaccination". Pharmacy staff who practice in our partnered independent Western Washington State community pharmacies will be eligible for this study. We plan to use the information we learn from the study to create a process that facilitates HPV and other adolescent vaccinations in pharmacies.

We are reaching out to you because you work at one of the pharmacies who has partnered with us on this study. Your decision to participate in this research study is voluntary. You do not have to participate if you do not wish to do so.

#### If you choose to participate in this 3-5-month study, you will be asked to:

- Review this consent form, ask study staff to answer any questions you have, and click on the "I Consent" button below if you decide to participate in the study.
- Complete two, 10–15-minute, online surveys. The first survey will begin following your
  decision to click on the "I Consent" button below. The second survey will be at the end of
  the study. Our goal is to collect pre/post surveys from up to 25 pharmacy staff members
  from the participating pharmacies.
- Attend two (2) 60-minute training session explaining a new communication strategy. The
  first session will be online provided as pre-recorded continuing education provided through
  the Washington State Pharmacy Association (WSPA). The second session will be live, in
  person or conducted online using Zoom, and will also count as CE administered through
  WSPA.
- Employ the new communication strategy for HPV vaccinations for 3 to 5 months.
- Designated pharmacy staff members will keep track of the following de-identified data:
   Age, sex/gender, race/ethnicity (if captured), insurance status, vaccine type, pharmacy
   where the patient was immunized, pharmacist who immunized the patient (using a unique
   code assigned to each pharmacist) for the duration of the intervention.

#### V. 11/10/2022 CTMS# RG1007825, IR# 10600

### PROMOTE Pilot Study Pharmacy Staff Aim 2 Online Consent Form

Your participation is voluntary. You can stop or withdraw from the study at any time or refuse to answer any questions. Employment of pharmacy staff will not be affected if staff either wish or do not wish to participate in this study.

All data collected will remain confidential. Information you share during the training session and pre and post intervention surveys will remain private. It will be stored without identifying information to protect your confidentiality. Study results will be published in aggregate.

Research is designed to benefit society by gaining new knowledge. You may not benefit personally from participating in the study. We anticipate few risks or discomforts involved from participating in this quality improvement study.

Participants will receive \$40 cash for completing both surveys to thank them for their time.

This study is being funded by the National Cancer Institute and has been approved by the Fred Hutchinson Cancer Center Institutional Review Board (IRB).

Some people or organizations may need to look at your research records for quality assurance or data analysis. They include:

- · Researchers involved with this study.
- Fred Hutchinson Cancer Center and its agents.
- Fred Hutchinson Cancer Center Institutional Review Board (IRB). An IRB is a group that reviews the study to protect your rights as a research participant.
- Office for Human Research Protections, and other agencies as required.

If you have questions about this study, please contact Dr. Parth Shah. His contact information is below.

If you have questions about your rights as a research participant in general, you may contact the Director of the Fred Hutch Institutional Review Office at <a href="mailto:irodirector@fredhutch.org">irodirector@fredhutch.org</a> or 206-667-5900.

Please click on the "I Consent" button below if you agree to participate in this study.

Thank you very much for your consideration.

Sincerely,

Parth Shah, PharmD, PhD (Primary Investigator)

### V. 11/10/2022 CTMS# RG1007825, IR# 10600

# PROMOTE Pilot Study Pharmacy Staff Aim 2 Online Consent Form

**Assistant Professor** 

Hutchinson Institute for Cancer Outcomes Research, Fred Hutchinson Cancer Center 1100 Fairview Ave. N., MS: M3-B232

Seattle, WA 98109

Office: 206-667-6120 Email: promote@fredhutch.org or pshah@fredhutch.org

I Consent